CLINICAL TRIAL: NCT04268381
Title: Local And Systemic Levels of aMMP-8 in Gingivitis and Stage 3 Periodontitis
Brief Title: Oral and Systemic aMMP-8 in Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Giresun University (Other)
Responsible Party: Principal Investigator, Zeynep Pinar KELES YUCEL, Assistant Prof., Giresun University
Other Study IDs: 20-2T/39
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Periodontal Diseases; Periodontal Inflammation
Keywords: periodontitis; gingivitis; matrix metalloproteinases
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy (n=23)
  Interventions: Other: Biochemical analysis
- Gingivitis (n=20)
  Interventions: Other: Biochemical analysis
- Periodontitis (n=40)
  Interventions: Other: Biochemical analysis

INTERVENTIONS:
Other: Biochemical analysis — aMMP-8 is measured by immunofluorometric assay (IFMA).

SUMMARY:
Periodontal disease is an inflammatory process that can result in tooth loss and also is considered a modifying factor for systemic health. Matrix metalloproteinase (MMP)-8 is the major collagenase of periodontal tissue breakdown. The aim of the present study is to analyze active (aMMP-8) levels in gingival crevicular fluid (GCF), saliva and serum in the context of new criteria of gingivitis and stage 3 grade C periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy and non-smoker individuals aged 25 to 50 years
* having ≥20 teeth present (except third molars)
* individuals with periodontally healthy, gingivitis and stage 3 periodontitis diagnoses

Exclusion Criteria:

* having any systemic disease
* smoking
* pregnancy or lactation
* using antibiotic or any anti-inflammatory drug or any periodontal treatment within the past 6 months.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy controls (n=23) includes volunteers with clinically healthy periodontium who had BOP < 10% and PD ≤ 3 mm, no sites with > 1 mm attachment loss, no radiographic sign of alveolar bone destruction and no history of periodontitis. Gingivitis patients (n=20) shows PD ≤ 3 mm with BOP > 50% in the entire mouth as well as no clinical attachment loss or alveolar bone loss. Periodontitis patients (Generalized Stage 3) have interdental CAL ≥ 5 mm at least 2 non-adjacent teeth, PD ≥ 6 mm and radiographic bone loss affecting 30% of the teeth or more.They show also no more than 4 teeth loss due to periodontitis.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Oral (GCF and saliva) and serum levels of aMMP-8 in periodontitis and gingivitis | through study completion, an average of 4 months
  aMMP-8 levels

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Pinar Keles Yucel, Principal Investigator — Department of Periodontology, School of Dentistry, Giresun University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No